CLINICAL TRIAL: NCT05633654
Title: A Randomized, Open-label, Phase 3 Study of Adjuvant Sacituzumab Govitecan and Pembrolizumab Versus Treatment of Physician's Choice in Patients With Triple Negative Breast Cancer Who Have Residual Invasive Disease After Surgery and Neoadjuvant Therapy
Brief Title: Study of Sacituzumab Govitecan-hziy and Pembrolizumab Versus Treatment of Physician's Choice in Patients With Triple Negative Breast Cancer Who Have Residual Invasive Disease After Surgery and Neoadjuvant Therapy (ASCENT-05/AFT-65 OptimICE-RD/GBG 119/NSABP B-63)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Alliance Foundation Trials, LLC. (Other); NSABP Foundation Inc (Network); GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-595-6184; 2024-512279-10 (Other: European Medicines Agency)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
Keywords: AFT-65; GBG 119; NSABP B-63; OptimICE-RD
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; pembrolizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab govitecan-hziy (SG) + Pembrolizumab (Experimental): Participants will receive SG 10 mg/kg intravenously on Days 1 and 8 of 21-day cycles and pembrolizumab 200 mg intravenously on Day 1 of 21-day cycles for 8 cycles.
  Treatment will be administered until a maximum of 8 cycles, local or distant disease recurrence, unacceptable toxicity, physician decision, consent withdrawal, or death.
  Interventions: Drug: Sacituzumab govitecan-hziy (SG); Drug: Pembrolizumab
- Treatment of Physician's Choice (TPC): Pembrolizumab or Pembrolizumab + Capecitabine (Active Comparator): Participants will receive one of the following TPC regimens determined prior to randomization:
  * Pembrolizumab 200 mg intravenously on Day 1 of 21-day cycles for 8 cycles OR
  * Pembrolizumab 200 mg intravenously on Day 1 of 21-day cycles and capecitabine 1000 mg/m^2 orally twice daily on Days 1 through 14 of 21-day cycles for 8 cycles.
  Treatment will be administered until a maximum of 8 cycles, local or distant disease recurrence, unacceptable toxicity, physician decision, consent withdrawal, or death.
  Interventions: Drug: Pembrolizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Sacituzumab govitecan-hziy (SG) — Administered intravenously
  Other Names: GS-0132; IMMU-132; Trodelvy™
  Arms: Sacituzumab govitecan-hziy (SG) + Pembrolizumab
Drug: Pembrolizumab — Administered intravenously
  Other Names: KEYTRUDA®
Drug: Capecitabine — Tablets administered orally
  Other Names: Xeloda
  Arms: Treatment of Physician's Choice (TPC): Pembrolizumab or Pembrolizumab + Capecitabine

SUMMARY:
The goal of this study is to find out if the experimental product, sacituzumab govitecan-hziy (SG) in combination with pembrolizumab given after surgery, is effective and safe compared to the treatment of physician's choice (TPC) which includes either pembrolizumab or pembrolizumab plus capecitabine in participants with triple negative breast cancer that still remains after surgery and pre-surgical treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Age > 18 years, with residual invasive triple negative breast cancer (TNBC) in the breast or lymph nodes after neoadjuvant therapy and surgery:

  * TNBC criteria for the study is defined as estrogen receptor (ER) and progesterone receptor (PR) ≤ 10%, human epidermal growth factor receptor 2 (HER2)-negative per American Society of Clinical Oncology and College of American Pathologists (ASCO/CAP) guidelines (immunohistochemistry (IHC) and/or in situ hybridization (ISH)).
* Adequate excision and surgical removal of all clinically evident of disease in the breast and/or lymph nodes and have adequately recovered from surgery.
* Submission of both pre-neoadjuvant treatment diagnostic biopsy and resected residual invasive disease tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Individuals must have received appropriate radiotherapy and have recovered prior to starting study treatment.
* Adequate organ function.

Key Exclusion Criteria:

* Stage IV (metastatic) breast cancer as well as history of any prior (ipsi- or contralateral) invasive breast cancer.
* Prior treatment with another stimulatory or coinhibitory T-cell receptor agent (eg, cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), OX-40, cluster of differentiation 137 (CD137), prior treatment with any HER2-directed agent, prior endocrine therapy for > 4 weeks or planned concurrent endocrine therapy while receiving on-study treatment.
* Evidence of recurrent disease following preoperative therapy and surgery.
* Prior treatment with topoisomerase 1 inhibitors or antibody-drug conjugates (ADCs) containing a topoisomerase inhibitor.
* Individuals with germline breast cancer gene (BRCA) mutations.
* Myocardial infarction or unstable angina pectoris within 6 months of enrollment or history of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias or Left ventricular ejection fraction (LVEF) of < 50%
* Active serious infections requiring anti-microbial therapy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1514 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (iDFS) | Up to 60 months
  iDFS is defined as the time from the date of randomization to death from any cause or one of the following events (whichever occurs first): invasive local, regional, or distant recurrence, invasive contralateral breast cancer.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 96 months
  OS is defined as the time from the date of randomization until death due to any cause.
Distant Disease-free Survival (dDFS) | Up to 60 months
  dDFS is defined as the time from the date of randomization to death from any cause or one of the following events (whichever occurs first): distant recurrence, or second primary invasive cancer.
Recurrence-free Survival (RFS) | Up to 60 months
  RFS is defined as the time from the date of randomization to death from any cause or one of the following events (whichever occurs first): invasive local, regional, or distant recurrence.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 38 months plus 30 days
Percentage of Participants Experiencing Laboratory Abnormalities | First dose date up to 38 months plus 30 days
Time to Worsening (TTW) of Quality of Life (QoL) Based on Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B) Trial Outcome Index (TOI) Scores | Up to 60 months
  TTW of FACT-B TOI scores will be analyzed for each index, the TTW of FACT-B scores will be measured from the randomization date and to the time the participants first experienced a first score of worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (287):
- United States (180):
  - Alabama Oncology, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Arizona Oncology Associates, Prescott Valley, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Community Cancer Institute, Clovis, California
  - PIH Health Whittier Hospital, Downey, California
  - Compassionate Cancer Care Medical Group - Inc, Fountain Valley, California
  - Los Angeles Cancer Network, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Cancer at Beverly Hills, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Emad Ibrahim, MD, INC, Redlands, California
  - Sutter Institute for Medical Research, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Stockton Hematology Oncology Medical Group, Stockton, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Norwalk Hospital, Danbury, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital - Bay Care, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Midland Florida Clinical Research Center, L, Orange City, Florida
  - Orlando Health, Orlando, Florida
  - Cancer Care Centers of Brevard, Inc, Palm Bay, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Sacred Heart Medical Oncology Group, Pensacola, Florida
  - Sylvester Comprehensive Cancer Center, Plantation, Florida
  - Cleveland Clinic Florida, Martin North Hospital, Stuart, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Weston Hospital, Weston, Florida
  - University Cancer & Blood Center, LLC., Athens, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Pearlman Cancer Center, Valdosta, Georgia
  - St Lukes Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Health, Coeur d'Alene, Idaho
  - Northwestern Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University Healthsystem, Evanston, Illinois
  - Edward Hospital, Naperville, Illinois
  - West Suburban Medical Center- River Forest, River Forest, Illinois
  - Edward H. Kaplan MD & Associates - Hematology/Oncology of the North Shore, Skokie, Illinois
  - Springfield Clinic LLP, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - IU Health Arnett Hospital, Lafayette, Indiana
  - Franciscan Health Munster, Munster, Indiana
  - Mercy Medical Center, Cedar Rapids, Iowa
  - Mission Cancer & Blood - John Stoddard Cancer Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Mercy Health, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - Sinai Hospital of Baltimore, Inc., Baltimore, Maryland
  - St. Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins Medicine - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Medstar Franklin Square Medical Center, Baltimore, Maryland
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - James M Stockman Cancer Institute, Frederick, Maryland
  - Greater Baltimore Medical Center, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institude at Merrimack Valley, Methuen, Massachusetts
  - Dana Farber Cancer Institute @ Milford Regional Hospital, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center (DF/BWCC) in Clinical Affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Baystate Medical Center Inc., Springfield, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Ascension, Grosse Pointe Woods, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Ascension Providence Hospital Southfield Cancer Center, Southfield, Michigan
  - Trinity Health St. Joseph Mercy Ann Arbor, Ypsilanti, Michigan
  - Minnesota Oncology Hematology, PA, Maplewood, Minnesota
  - Virginia Piper Cancer Center (Allina Health), Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Baptist Clinical Research Institute, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Mary Lanning Healthcare - Morrison Cancer Center, Hastings, Nebraska
  - Oncology Hematology West - Methodist, Omaha, Nebraska
  - Nebraska Methodist Hospital (change from Chi Health Bergan Mercy), Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Cancer Care & Hematology Specialists, Reno, Nevada
  - Regional Cancer Care Associates LLC, East Brunswick, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Summit Medical Group, P.A., Florham Park, New Jersey
  - Rutgers Health, New Brunswick, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - San Juan Oncology Associates, Farmington, New Mexico
  - New York Oncology Hematology (NYOH), Amsterdam, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York, PC, East Syracuse, New York
  - Northwell Health, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Canter, New York, New York
  - Lipson Cancer Institute - Linden Oaks, Rochester, New York
  - New York Cancer and Blood Specialists, Shirley, New York
  - Stony Brook Medicine, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinical Research Alliance, Westbury, New York
  - White Plains Hospital Physician Associates, White Plains, New York
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Cone Health Medical Group (Moses Cone Health System), Greensboro, North Carolina
  - East Carolina University Health Medical Center, Greenville, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - UNC Rex Cancer Center, Raleigh, North Carolina
  - UNC Nash Cancer Center, Rocky Mount, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Columbus NCORP, Columbus, Ohio
  - Anita Stewart Oncology Center, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. Charles Health System, Inc. DBA St. Charles Medical Center, Bend, Oregon
  - Samaritan Hospital, Corvallis, Oregon
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Cancer Institute - Oncology Clinical Trials, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Saint Luke's University Hospital, Bethlehem, Pennsylvania
  - Lancaster General Health, Lancaster, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Providence Health, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Monument Health Cancer Care Institute, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Center for Biomedical Research, LLC, Knoxville, Tennessee
  - University of Tennessee, Knoxville, Tennessee
  - Hendrick Health System, Abilene, Texas
  - Texas Oncology, Austin, Texas
  - Texas Oncology, El Paso, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc, Wytheville, Virginia
  - Providence Regional Cancer System, Lacey, Washington
  - MultiCare Regional Cancer Center - Tacoma, Puyallup, Washington
  - Northwest Medical Specialties, PLLC, Puyallup, Washington
  - University of Washington, Renton, Washington
  - Medical Oncology Associates, Spokane, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension St. Francis Reiman Cancer Center, Franklin, Wisconsin
  - HSHS Saint Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Australia (6):
  - Macarthur Cancer Therapy Centre, Campbelltown Hospital, Campbelltown, New South Wales
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- France (13):
  - CHU Amiens Picardie, Amiens
  - Pôle Santé Léonard De Vinci - ROC37, Chambray-lès-Tours
  - Clinique Victor Hugo, Le Mans
  - chu de Limoges, Limoges
  - Hôpital Privé Jean Mermoz, Lyon
  - Centre D'Oncologie de Gentilly, Nancy
  - L'Hôpital Privé du Confluent, Nantes
  - CHU de Nimes, Nîmes
  - Hopital Privé des Côtes d'Armor - Centre CARIO-HPCA, Plérin
  - CHU de Poitiers, 2 Rue de la Milétrie, Poitiers
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest (ICO) - St Herblain, Saint-Herblain
  - Oncopole Claudius Regaud - IUCT-O, Toulouse
- Germany (42):
  - Hämatologie-Onkologie im Zentrum MVZ GmbH, Augsburg
  - Schwanebecker Chaussee 50, Berlin
  - Möllendorffstr. 52, 10367 Berlin 2. Behandlungsstandort: Markt 2-3, 13597 Berlin, Berlin
  - Teutoburger Str. 60, Bielefeld
  - Josef-Albers-Str.70, Bottrop
  - Studien GbR Braunschweig, Braunschweig
  - St.-Juergen-Str. 1, Bremen
  - Hämato-Onkologische Praxis im Medicum, Bremen
  - St. Elisabeth Krankenhaus GmbH, Cologne
  - St. Johannes Hospital, Dortmund
  - Fetscherstraße ,74, Dresden
  - Klinikum Essen-Mitte, Düsseldorf
  - Henricistraße 92, 45136 Essen, Germany, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Wilhelm-Epstein-Str. 4, Frankfurt
  - Gotenstraße 6-8, Frankfurt am Main
  - Hugstetter Str. 55, Freiburg im Breisgau
  - Munckelstrasse 27, Gelsenkirchen
  - MVZ II der Niels Stensen Kliniken, Georgsmarienhütte
  - Straße des Friedens 122, Gera
  - Moorkamp 2-6, Hamburg
  - Am Klinikum 1, Jena
  - Edgar-von-Gierke-Straße 2, Karlsruhe
  - Elisabeth Krankenhaus Brustzentrum, Kassel
  - InVO - Institut für Versorgungsforschung in der Onkologie GbR / Praxis für Hämatologie und Onkologie, Koblenz
  - Fachärztezentrum Langen, Langen
  - Biedermannstrasse 84, Leipzig
  - Universitätsklinikum Mannheim, Mannheim
  - Taxisstrasse 3, Munich
  - Bei der Marienkirche 6, Mühlhausen
  - Albert-Schweitzer-Campus 1, Building A1,, Münster
  - Charlottenstraße 72, Potsdam
  - Elisabethenstr. 19, 88212 Ravensburg, Ravensburg
  - Südring 81, Rostock
  - Harsefelderstraße 8, Stade
  - Böheimstr. 37, Stuttgart
  - Schierghoferstrasse 1, Traunstrein
  - Calwerstrasse 7, Tübingen
  - Prittwitzstr. 43, Ulm
  - Beethovenstrasse 20, Wiesbaden
  - Klinikum Worms Frauenklinik, Worms
  - Helios University Hospital University Witten/Herdecke, Wuppertal
- Ireland (5):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Limerick, Limerick
- South Korea (5):
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (34):
  - Medical Oncology Unit. A Coruña University Hospital, A Coruña
  - ICO Badalona - Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitary of Cruces, Barakaldo
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castellon
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital Reina Sofia, Córdoba
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital General Universitario De Elche, Elche
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Galdakao, Galdakao
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario de Jaen, Jaén
  - H. León, León
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Beata María Ana, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Althaia Xarxa Assistencial de Manresa, Manresa
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hosp. Mat-Inf. Carlos Haya, Málaga
  - Hospital General Univers, Murcia
  - Hospital Universitario Morales Meseguer, Murcia
  - Clínica Universidad de Navarra - Madrid, Pamplona
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - HU Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quironsalud Sagrado Corazón, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Isabel la Catolica nº 1-3, Zaragoza
- United Kingdom (2):
  - Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tolaney SM, DeMichele A, Takano T, Rugo HS, Perou C, Lynce F, Parsons HA, Santa-Maria CA, Rocque GB, Yao W, Sun SW, Mocci S, Partridge AH, Carey LA. OptimICE-RD: sacituzumab govitecan + pembrolizumab vs pembrolizumab (+/- capecitabine) for residual triple-negative breast cancer. Future Oncol. 2024;20(31):2343-2355. doi: 10.1080/14796694.2024.2357534. Epub 2024 Jun 26. PMID 38922307
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-595-6184